CLINICAL TRIAL: NCT04147000
Title: Pharmacokinetics and Pharmacodynamics of Oral Sertraline Before and After Bariatric Surgery; a Prospective Open Observational Study
Brief Title: Pharmacokinetics and Pharmacodynamics of Oral Sertraline Before and After Bariatric Surgery
Acronym: ANTILOP
Status: Terminated | Type: Observational
Why Stopped: Problem with recruiting as a consequence of COVID-19
Sponsor: Linkoeping University (Other Government)
Collaborators: Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Michael Andresen, Principal Investigator, Linkoeping University
Other Study IDs: ANTILOP
Record Dates: First submitted 2019-10-28; First posted 2019-10-31 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Overweight; Depression; Anxiety Disorders
Keywords: Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Overweight; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum from blood samples, frozen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Volunteers with a prescription of oral sertraline who have been scheduled to bariatric surgery in either Norrköping/Sweden or Lindesberg/Sweden will be asked to participate in a observational study. The aim of this study is to evaluate the absorption and the effect and side effects of sertraline in volunteers 8 weeks before and 1, 6 and 12 months after bariatric surgery.

DETAILED DESCRIPTION:
The pharmacokinetic changes of sertraline after bariatric surgery are studied by assessing the exposition for sertraline in individuals with long term treatment by measuring the area under the curve (AUC0-τ) 8 weeks before and one, six and twelve months after bariatric surgery in 30 participants.

The effect of variation of sertraline concentration is studied by a psychiatric assessment of depressive symptoms and symptoms of anxiety disorder. The aim ist to study if there is a relation between changes in pharmacokinetics and effect of sertraline after bariatric surgery.

For the assessment of side effects a self-reporting scale is used. These participants are recruited consequentially with the aim to get equal numbers of patients with both most usual types of surgery in Sweden (laparoscopic RYGB and gastric sleeve).

ELIGIBILITY:
Inclusion Criteria:

* scheduled to undergo either gastric bypass or gastric sleeve surgery via surgeon clinics in Örebro or Norrköping
* prescription of sertraline
* since at least one month
* planned to be continued at the time of inclusion
* swedish speaking

Exclusion Criteria:

* comorbidity with the consequence that the potential participant may not be able to complete the study
* if participation should result in a high risk for patients health or safety

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Volunteers scheduled for bariatric surgery in one of the two participating surgical clinics. Consecutive sampling until 30 volunteers are recruited.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-11-12 (Actual); Study Completion 2023-11-12 (Actual)

PRIMARY OUTCOMES:
Change in Area under the concentration curve of sertraline | 8 weeks before, 1, 6 and 12 month after bariatric surgery before sertraline intake and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8 and 24 hours post dose
  Changes in the area under sertraline serum concentration vs time curve (AUC(0-t))
Change in Clinical Anxiety Scale | 8 weeks before, 1, 6 and 12 month after bariatric surgery
  Psychiatric assessment of symptoms of anxiety disorders with an 5-items-scale (Psychic tension, Ability to relax/muscular tension, Startle response/hyperarousability, Worrying, Apprehension). Every item has values between 0 (no symptoms) and 4 (marked symptoms). The overall score ranges from 0 to 20.Higher scores indicate higher anxiety symptoms.
Change in Montgomery-Åsberg-depression rating scale (MADRS-B) | 8 weeks before, 1, 6 and 12 month after bariatric surgery
  Assessment of depressive symptoms with a 10-items scale (Apparent Sadness, Reported Sadness, Inner Tension, Reduced Sleep, Reduced Appetite, Concentration Difficulties, Lassitude, Inability to Feel, Pessimistic Thoughts, Suicidal Thoughts). Higher score indicates more depressive symptoms, each item spans over a score from 0 to 6; the overall score ranges from 0 to 60.

SECONDARY OUTCOMES:
Changes in the area under concentration vs time curve of desmethylsertraline | 8 weeks before, 1, 6 and 12 month after bariatric surgerybefore sertraline intake and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8 and 24 hours post dose
  Changes in the area under concentration vs time curve of desmethylsertraline

CONTACTS AND LOCATIONS:
Overall Officials: Michael Andresen, MD, Principal Investigator — Linkoping university, Örebro university; Ylva Böttiger, Professor, Study Director — Linkoeping University
Locations (2):
- Sweden (2):
  - Lindesbergs lasarett, Lindesberg, Örebro County
  - Vrinnevisjukhus, Norrköping, Östergötland County

IPD SHARING:
Plan to Share IPD: No